CLINICAL TRIAL: NCT02475980
Title: Providing Adolescent Contraception in the Emergency Room (PACER)
Brief Title: Providing Adolescent Contraception in the Emergency Room
Acronym: PACER
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Other Study IDs: 14-248; 3RX15 (Other Grant/Funding Number: Society of Family Planning)
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Contraception
Keywords: Adolescent; Contraception; Counseling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescent girls: Adolescent post-menarchal girls ages 13-18 with Medicaid insurance presenting to a pediatric emergency department for a non-emergent complaint who receive comprehensive contraception counseling
  Interventions: Behavioral: Comprehensive contraception counseling

INTERVENTIONS:
Behavioral: Comprehensive contraception counseling — The study intervention will consist of comprehensive contraceptive counseling through a standardized bundle of services, including a 10-minute educational DVD, handouts on contraceptive methods, and one-on-one contraceptive counseling by the PED physician.

SUMMARY:
The purpose of this pilot study is to determine the feasibility of comprehensive contraceptive counseling intervention in a pediatric emergency department and to determine the impact of comprehensive contraception counseling on initiation of contraception among sexually active adolescents presenting to a pediatric emergency department.

DETAILED DESCRIPTION:
Adolescent pregnancy is a crippling problem. Despite declines in adolescent birth rates, adolescent pregnancies cost taxpayers a staggering $9.4 billion in 2010. New Mexico has one of the highest rates of adolescent pregnancy in the country.(1) In New Mexico, nearly 1 in 5 adolescent females are not using any form of contraception.(2) Long-acting reversible forms of contraception, including the subdermal contraceptive implant known as Nexplanon, are increasingly popular among adolescents. Nonetheless, despite an increase from 0.3% in 2000 to 4.5% in 2013, few adolescents using any contraception are using a long-acting reversible form.(1) The American College of Obstetricians and Gynecologists issued a policy statement in late 2012 recommending long-acting, reversible forms of contraception as first line contraception for adolescents.(3) Long-acting, reversible forms of contraception are highly effective at preventing pregnancy and have rates of continuation among adolescents comparable to older women.(4) Prior studies of adolescents have demonstrated that cost, access, and education are the primary barriers to initiation of long-acting reversible forms of contraception and that, if these barriers are removed, acceptance rates approach 75%.(5,6) However, adolescents at highest risk of pregnancy have few opportunities to obtain highly-effective contraception.

The contribution of the proposed research is to demonstrate the feasibility of providing comprehensive counseling about contraception for adolescents in a novel outreach setting, a pediatric emergency department. This contribution will be significant because, if this counseling intervention increases initiation of contraception through a pediatric emergency department, unintended pregnancies among vulnerable adolescents may decrease. The term vulnerable will be used throughout this application to refer to adolescent girls who seek care for non-emergent complaints in emergency departments, are likely to be publicly insured or uninsured, engage in risky behaviors, have co-morbid psychiatric disorders, or have high-risk social characteristics such as interpersonal violence, substance abuse, or poverty.(7-9) Vulnerable adolescents are at high risk of unintended pregnancy, yet are difficult to reach through outpatient care settings. Initiation of contraception at the time of pediatric emergency department encounter could reduce unintended pregnancy, reduce adverse outcomes to the woman and her child associated with adolescent pregnancy, and reduce the financial costs borne by society.

Currently, most contraception for adolescents is initiated through an outpatient encounter. In New Mexico, adolescent girls aged 13 to 18 who present to an outpatient clinic for contraception can be prescribed contraception or have a contraceptive device placed during the clinic visit without parental consent under state law.(10) This approach has enjoyed considerable success, with a 15-fold increase in the use of intrauterine or subdermal contraceptive implants by adolescents seeking contraception over the past decade.(1) The Contraceptive CHOICE study has demonstrated that adolescents have high acceptance of long-acting, reversible forms of contraception.(5) Typically, providers of highly-effective contraception are gynecologists, advanced practice physicians, and family practice physicians. This has resulted in a scarcity of providers who can offer the long-acting, reversible contraception to adolescents that is recommended by the American College of Obstetricians and Gynecologists.(3,11) Additionally, not all adolescents are able to access clinic-based, outpatient medical care by a gynecologist or family practitioner. Adolescents who experience poverty, coercive sexual relationships, co-morbid psychiatric disorders, and abuse are especially vulnerable to pregnancy.(12) These risk factors for adolescent pregnancy mirror the characteristics of adolescents who utilize emergency departments for medical care.(7-9,13) A prior survey of female adolescents and adults seeking care in an emergency department felt it was acceptable to have contraceptive provision in the emergency department. (14)

It is not known whether pediatric emergency medical providers can successfully initiate contraception for adolescents in a pediatric emergency department. Adolescent girls who present to the UNM Pediatric Emergency Department (PED) currently receive some contraceptive and sexual health care, but the care delivered varies based on the provider.

As a continuing education initiative at UNM, Dr. Nancy Sokkary, Adolescent Gynecologist, has been providing educational sessions on current best contraceptive practices for adolescents to pediatricians. Included in this education has been an FDA-approved procedural training in the insertion of the subdermal contraceptive implant, Nexplanon. Pediatric residents and attending physicians have begun to offer Nexplanon in the inpatient setting and in pediatric clinics. As PED attending and fellow physicians, all of whom are board-certified pediatricians, undergo this education, we anticipate increased knowledge on the part of PED providers on current contraceptive recommendations. This proposed research capitalizes on an opportunity to expand comprehensive counseling on contraception in the PED.

Patients will be recruited through the Pediatric Emergency Department (PED) of the University of New Mexico. Investigators will enroll adolescent girls 13 to 18 years of age who present to the PED for non-emergent complaints and who are willing to participate in the study. Adolescent girls who present to the PED during shifts staffed by an attending physician or fellow trained in the study counseling intervention will be eligible for enrollment. Physicians who have completed Dr. Sokkary's continuing education on best practices in adolescent contraception and the FDA-approved Nexplanon insertion training will be considered trained in the counseling intervention. All consents and procedures will be performed in the PED by a research coordinator or study investigator who will not be involved in the patient's medical care during their emergency department encounter. All potentially eligible participants will be approached by the research coordinator while their parent/guardian/companion is outside of the patient room, as is routine for reproductive health care in the PED. A unique study number will be assigned to each subject and noted on all data collection forms containing only the study number. No patient identifiers will be included on the data forms.

All patients will be offered clinical services regardless of their decision about participating in the study. If a participant is withdrawn from the study either by her desire or that of the PED provider, the PI of the study or the research staff, she may continue to receive contraceptive care which will be up to the PED clinician providing clinical services during the encounter.

Patients can expect that participation will involve enrollment and a subsequent contraceptive counseling intervention consisting of a handout, 10-minute DVD, and a one-on-one counseling by a PED attending physician or fellow that will not total longer than one hour. For follow up, all participants will be contacted by telephone by a study team member approximately 4 weeks after enrollment and will be administered a brief (approximately 10 minute) survey on participant satisfaction with the counseling intervention and on any subsequent contraceptive choices. Investigators will recruit participants during an 8-week pilot period. Investigators anticipate recruitment to be completed by March of 2015 and preliminary analysis to be complete by June 2015.

Participants will be recruited through the Pediatric Emergency Department (PED) at UNM. Physicians in the Pediatric Emergency Department (PED) are trained Pediatricians who provide specialized care in Emergency Medicine. Sixty percent of PED attendings and fellows completed training by Dr. Sokkary on best practices in adolescent contraception and in Nexplanon insertion during September 2014.

Usual care for contraceptive counseling in the PED:

The most common reason that adolescent girls present to the PED is persistent abdominal pain. Other common reasons include urinary tract infections, concern for sexually transmitted infections, pharyngitis, upper respiratory tract infections, social stressors, and trauma. An adolescent girl's first point of care in the PED is nurse triage. PED visits by adolescent girls average a total duration of just over 4 hours. During nurse triage, a brief history of the presenting complaint is taken, vital signs are collected, and medical care is initiated based on nurse-driven protocols. During triage, female adolescent patients are routinely interviewed privately with parent/guardian/companion outside of the room to screen for pregnancy risk factors. They are provided with a urine specimen cup in anticipation of urine pregnancy testing. Depending on the chief complaint, the triage nurse may privately screen for other risk factors such as substance abuse or violence. After triage, the patient is placed in one of 12 private patient rooms in the PED. They are evaluated by one to three physicians in the PED depending on the staffing of the PED at that time. Medical evaluation routinely consists of a medical history and a physical exam. In addition, routine care of adolescents in the PED includes a social history that is obtained with the parent/guardian/companion outside of the patient's room to protect confidentiality. During the confidential portion of the medical encounter, most adolescents are asked about sexual behavior, contraception, healthy relationships, and substance abuse. Currently, PED providers offer contraceptive counseling on a case-by-case basis. If contraception counseling is included as part of the confidential medical encounter, this is not a deviation from routine care that the adolescent would receive in an outpatient clinic visit for simple chief complaints. If adolescents express interest in initiating contraception or changing contraceptive methods, PED providers are able to offer a range of contraceptive services. The range of contraceptive services available in the PED include:

* Emergency contraception (given in PED or as prescription);
* Prescription for contraception (including oral contraceptive pills, vaginal ring, dermal patch);
* Immediate Depo-Provera injection;
* Immediate subdermal contraceptive implant insertion (only available if patient seen by a Nexplanon-trained provider); or,
* Referral to Adolescent Gynecology or Center for Reproductive Health for outpatient initiation of contraception, including the IUD or subdermal contraceptive implant.

Patients receiving contraceptive services in the PED are offered follow-up in Adolescent Gynecology as an outpatient as usual care.

The proposed research is a pilot study of a contraceptive counselling intervention, administered by Pediatric Emergency Medicine providers for adolescent girls presenting to the University of New Mexico Pediatric Emergency Department for non-contraceptive complaints. The primary research question is: Is it feasible to initiate comprehensive contraceptive counseling in a pediatric emergency department? The secondary research question is: What is the impact of comprehensive contraceptive counseling on the initiation of contraception among sexually active adolescents presenting to a pediatric emergency department?

The overall study design is a prospective cohort study. The two specific aims for the proposed research reflect the two key perspectives of stakeholders in this proposed pilot study. Specific aim #1, Determine the feasibility of comprehensive contraception counseling in a pediatric emergency department, investigates the introduction of a contraceptive practice within the existing time and resource constraints of emergency medical providers in a busy emergency department. Specific aim #2, Determine the impact of comprehensive contraceptive counseling on initiation of contraception among sexually active adolescents presenting to a pediatric emergency department, elicits the effectiveness of providing contraceptive counseling during an emergency department encounter from the perspective of adolescents. Feasibility, as operationalized in this application, requires attainment of our measurable, hypothesized outcomes by both participating emergency medical providers and adolescents.

Eligible participants will include post-menarchal girls ages 13 - 18 who present to the Pediatric Emergency Department for non-contraceptive complaints. Investigators will enroll subjects during an 8-week period. Subjects will only be enrolled during a patient care shift staffed by a Pediatric Emergency Medicine provider who has completed Dr. Nancy Sokkary's contraceptive educational session and Nexplanon insertion training as part of continuing education. Female adolescents will be screened for study eligibility at triage by a triage nurse using a standardized set of criteria (see Appendix A and B). The eligibility criteria include:

* Ages 13 to 18 years old
* Speaks English or Spanish
* Has menstrual periods
* Has Medicaid insurance
* Is not seeking contraception as their primary complaint
* Is not currently pregnant based on urine or serum pregnancy testing
* Does not have an IUD or contraceptive implant (Implanon/Nexplanon)
* Is not critically ill, hemodynamically unstable, altered mental status, developmentally delayed, severe pain or distress, or have major trauma

The triage nurse will alert the Unit Clerk who will contact the on-call research coordinator after verifying insurance eligibility criteria. The research coordinator will further determine study eligibility. Per usual care in the Pediatric ED, most adolescent girls will be screened for pregnancy by urine or serum testing as part of their routine medical care initiated through triage. A small number of adolescent girls may not be screened for pregnancy at triage or during their subsequent medical care according to usual care for their specific presenting complaints. If girls are otherwise eligible for study participation but have not undergone pregnancy testing as a routine part of their medical care in the PED, these potentially eligible participants will be provided with a point-of-care urine pregnancy test at no cost to the participant.

If patients are eligible and choose to participate in the research study, consent for participation will be obtained. Under the requested waiver of parental consent, potential participants will be consented and enrolled with the parents/guardian/companion outside of the patient's room. The research coordinator/study investigator will explain the constraints of confidentiality in accordance with the recruitment script (see Appendix C) and will explain that while reproductive health care is confidential, any disclosures of intent to self-harm, intent to harm others, or abuse perpetrated upon the participant will require immediate disclosure to the participant's PED medical provider. At the time of enrollment, the research coordinator/study investigator will administer a patient enrolment questionnaire that contains questions about demographics and factors that increase risk of adolescent pregnancy (Appendix D).

Data collection will be completed on the same day as the patient's emergency department encounter by the research coordinator/study investigator and stored using REDCap. The REDCap database will be stored on a secure server at the University of New Mexico Health Sciences Center (UNM HSC), and the database will only be accessed by University of New Mexico's Human Resources Protections Office (HRPO) approved co-investigators on UNM HSC password-protected computers. Patients will fill out contact information on paper collection forms and the information will then be entered into an Access database. Demographic characteristics and any questionnaires will be collected on paper forms and entered into the REDCap database. All data will be destroyed 7 years after HRPO completion date with patient information destroyed via shredding of paper documents. Patient identifiers linked to the data will be destroyed by removal of the file from the hard drive of the UNM computer used to store the information.

The study intervention will consist of comprehensive contraceptive counseling through a standardized bundle of services, including a 10-minute educational DVD, handouts on contraceptive methods, and one-on-one contraceptive counseling by the PED physician. Patients who are enrolled in the study will have a color-coded tag applied to their physical patient chart and the door of their room at the time of enrollment. Emergency department ancillary staff will bring the educational DVD developed specifically for this project by UNM Family Planning and Adolescent Gynecology providers (see Appendix E) and the educational handouts (see Appendix F) to the room at the time that the tag is displayed. Every room in the PED is equipped with a combination DVD player/video display. All participating patients will also receive one-on-one contraceptive counseling by one the of Pediatric Emergency Medicine providers after watching the DVD.If study participants express interest to the PED provider in initiating contraception or changing to a more effective method of contraception after receiving the counseling intervention, participants will be offered all available options in the PED for which they are medically eligible as per usual care All participants will be contacted by telephone by a research coordinator approximately 4 weeks after enrollment and administered a questionnaire (see Appendix G) regarding their satisfaction with receiving contraceptive counseling in the Pediatric Emergency Department and any subsequent changes in their contraceptive practices. Additionally, all participants will undergo a one-time chart review at approximately 4 weeks post-enrollment to determine the rate of successful follow-up with Adolescent Gynecology or Center for Reproductive Health for this group.

At the end of the 8 week intervention, the Pediatric Emergency Medicine providers who participated in Dr.Sokkary's contraceptive educational session and the study intervention will complete a short survey (see Appendix I: Provider Questionnaire) administered by the research coordinator. This survey is to elicit the physicians' impressions regarding patient throughput during the clinical intervention, as well as impact on physician workflow. No personal or identifying information will be collected from the providers. We are requesting for a waiver of written documentation of consent for this PED provider survey.

This study will recruit adolescent girls presenting to the Pediatric Emergency Department. Adolescents who seek care for non-emergent complaints in emergency departments may be an especially vulnerable population, as prior research has demonstrated that these adolescents are likely to be publicly insured or uninsured, engage in risky behaviors, have co-morbid psychiatric disorders, or have high-risk social characteristics such as interpersonal violence, substance abuse, or poverty (Melzer-Lange, 1996; Wilson, 2000; Ziv, 1998). Adolescents who experience poverty, coercive sexual relationships, co-morbid psychiatric disorders, and abuse are especially vulnerable to pregnancy (Klein, 2005). These risk factors for adolescent pregnancy mirror the characteristics of adolescents who utilize emergency departments for medical care. Investigators hope to improve access to contraceptive care for this group of adolescents. However, to avoid coercion, no incentives for study participation will be offered. Because adolescents who seek care in emergency departments are more likely to have high-risk social characteristics, it is possible that participants may disclose physical or sexual abuse, assault, commercial sexual activity, suicidality, or homicidality. Any disclosures that qualify for mandated reporting that occur within the study will be disclosed immediately to the attending PED provider so that appropriate child safety authorities can be notified. Coordination of care with child safety authorities is routine care in the PED and child safety authorities, including CYFD and law enforcement agencies, are contacted by the PED daily in the course of routine care.

ELIGIBILITY:
Inclusion Criteria:

* Ages 13 to 18 years old
* Speaks English or Spanish
* Has menstrual periods
* Has Medicaid insurance

Exclusion Criteria:

* Seeking contraception as their primary complaint
* Currently pregnant based on urine or serum pregnancy testing
* Has an IUD or contraceptive implant (Implanon/Nexplanon)
* Critically ill, hemodynamically unstable, altered mental status, developmentally delayed, severe pain or distress, or have major trauma
* In juvenile justice custody

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent girls presenting to a pediatric emergency department for non-emergent complaints
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adolescent Girls
Started | 13
Completed | 8
Not Completed | 5
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adolescent Girls
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.85 (1.675)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay
Description: Emergency department length of stay for participants
Time Frame: Measured at time of chart review for patient follow-up, approximately 4 weeks after enrollment.
Measure: Median (Full Range); unit: minutes
Arm/Group | Adolescent Girls
Number analyzed (Participants) | 13
minutes | 287 [103 to 895]

2. Primary Outcome: Proportion of Eligible Girls Offered Counseling Intervention
Description: Proportion of girls eligible to participate in study who were offered contraceptive counseling
Time Frame: Approximately 4 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Adolescent Girls
Number analyzed (Participants) | 13
participants | 13

3. Primary Outcome: Participant Satisfaction
Description: Participant ratings of acceptability of contraceptive counseling in the emergency department and satisfaction with counseling
Time Frame: 4 weeks after enrollment
Population: Number of girls available for follow-up at 4-week phone call.
Measure: Number; unit: participants
Arm/Group | Adolescent Girls
Number analyzed (Participants) | 8
participants
  Reported Extremely Satisfied | 4
  Reported Somewhat Satisfied | 3
  Reported Neither satisfied nor dissatisfied | 1
  Reported Somewhat dissatisfied | 0
  Reported Extremely Dissatisfied | 0

4. Primary Outcome: Contraceptive Initiation
Description: Proportion of participants who report initiating contraception or changing to a more effective method of contraception
Time Frame: 4 weeks after enrollment
Population: Of the 13 girls consented to the study, 1 initiated a new contraception method following the intervention.
Measure: Number; unit: participants
Arm/Group | Adolescent Girls
Number analyzed (Participants) | 13
participants | 1

5. Secondary Outcome: Descriptive Statistics of Participants
Description: Frequencies and descriptive statistics of participant demographics, comorbidities associated with unintended adolescent pregnancy, and contraceptive use
Time Frame: At conclusion of study data collection, approximately 8 weeks after enrollment
Population: Participants consented for project
Measure: Number; unit: participants
Arm/Group | Adolescent Girls
Number analyzed (Participants) | 13
participants
  Reported unintended adolescent pregnancy | 2
  Reported a history of abortion | 1
  Reported having used a condom | 2
  Reported current use of non-LARC contraception | 5

6. Secondary Outcome: Follow-up Adherence
Description: Proportion of girls who present for follow-up appointment after referral to Adolescent Gynecology outpatient clinic
Time Frame: 4 weeks after enrollment
Population: Number of participants given a referral to Adolescent Gynecology in PED
Measure: Number; unit: participants
Arm/Group | Adolescent Girls
Number analyzed (Participants) | 5
participants
  Appointment not scheduled | 3
  Appointment scheduled | 2
  Presented to Adolescent Gynecology follow-up appt | 0

ADVERSE EVENTS:
Arm/Group | Adolescent Girls
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No